CLINICAL TRIAL: NCT01417702
Title: Advanced Endoscopic Imaging Using HD+ Endoscopy and i-Scan for Assessment of Mucosal Healing in IBD
Brief Title: Endoscopy for Assessment of Mucosal Healing in IBD
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: HN-0007
Record Dates: First submitted 2011-08-10; First posted 2011-08-16 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Crohn´s Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Crohn´s disease - active: Patients in the active phase of the disease
  Interventions: Device: High-definition white light endoscopy and i-Scan
- Crohn´s disease - quiescent: Patients in the quiescent phase of the disease
  Interventions: Device: High-definition white light endoscopy and i-Scan
- Ulcerative colitis - active: Patients in the active phase of the disease
  Interventions: Device: High-definition white light endoscopy and i-Scan
- Ucerative colitis - quiescent: Patients in the quiescent phase of the disease
  Interventions: Device: High-definition white light endoscopy and i-Scan

INTERVENTIONS:
Device: High-definition white light endoscopy and i-Scan — Patients will undergo advanced endoscopic imaging. Findings will be compared to histopathological and clinical results.

SUMMARY:
Inflammatory bowel disease (IBD) encompasses two major forms of chronic intestinal disorders, Crohn's disease and ulcerative colitis (UC). Diagnosis is based on several macroscopic and histologic features including patterns of inflammation, crypt abscesses and granulomas. i-Scan use an endoscopic image from the video processor and reconstruct virtual images in real time, resulting in an improved contrast of the capillary patterns and enhancement of the mucosal surface (so called virtual chromoendoscopy).

The main objective of this study is to determine endoscopic features of mucosal healing in patients with IBD and to compare these features to clinical and histological data in order to establish a new endoscopic classification of mucosal healing and to evaluate mucosal healing as a parameter of remission and relapse.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18-85 years
* Ability of subjects to understand character and individual consequences of clinical trial
* Subjects undergoing colonoscopy

Exclusion Criteria:

* Inability to provide written informed consent
* Severe Coagulopathy (Prothrombin time < 50% of control, Partial thromboplastin time > 50 s)
* Pregnancy or breast feeding
* Active gastrointestinal bleeding
* Residing in institutions (e.g. prison)
* Proctocolectomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn´s disease and ulcerative colitis were prospectively included.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Mucosal healing | up to three years
  We will determine high-definition white light endoscopic and i-Scan features of mucosal inflammation (e.g. erosions, erythema, ulcerous lesions) in IBD in order to establish a new endoscopic classification of mucosal healing.

SECONDARY OUTCOMES:
Histologic correlation | up to three years
  Comparison of clinical and histopathological data with endoscopic findings to evaluate mucosal healing as a parameter of remission and relapse.
Therapeutic effect | up to three years
  We will evaluate the effect of different therapeutic strategies (eg. anti-TNF treatment) on characteristics (e.g. erosions, ulcers, erythema) of mucosal healing.

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Neumann, Professor, Principal Investigator — Department of Medicine I, University of Erlangen-Nuremberg, Germany; Markus F. Neurath, Professor, Principal Investigator — Department of Medicine I, University of Erlangen-Nuremberg, Germany
Locations (1):
- University of Erlangen-Nuremberg, Erlangen, Germany